CLINICAL TRIAL: NCT02693782
Title: Effect of Wheat Bran Extract Containing Arabinoxylan Oligosaccharides, on the Gut Microbiota Composition and Well-being in Healthy Aging Subjects PhD Project: New Targeted Prebiotic Approaches for Maintaining Human Health
Brief Title: Fabulous Fibre Study - Effect of Wheat Bran Extract on Gut and General Health in Healthy Aging Subjects (FFS)
Acronym: FFS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Collaborators: Cargill (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 15/HSMC/004
Record Dates: First submitted 2015-06-29; First posted 2016-02-29 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2016-09

CONDITIONS: Hypercholesterolemia; Flatulence; Intestinal Diseases
Keywords: Fibre; Wheat Bran Extract; Microbiota; Microbiota metabolites; Gastrointestinal tolerance
MeSH Terms: conditions — Hypercholesterolemia; Flatulence; Intestinal Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): 15 g/day maltodextrin in 3 portions of 5 g.
  Interventions: Dietary Supplement: Placebo
- Fibre supplement (Active Comparator): 15 g/day Wheat Bran Extract in 3 portions of 5 g.
  Interventions: Dietary Supplement: Fibre supplement

INTERVENTIONS:
Dietary Supplement: Placebo — 15 g/day maltodextrin in 3 portions of 5 g.
  Arms: Placebo
Dietary Supplement: Fibre supplement — 15 g/day Wheat Bran Extract in 3 portions of 5 g.
  Arms: Fibre supplement

SUMMARY:
This is a placebo controlled, cross-over, randomized, double blinded study. The intervention food products will be taken as diet prebiotic supplements: 1. Wheat Bran Extract rich in arabinoxylan oligosaccharides : 15g/d (up to 10 g total additional dietary fibre per day). 2. Placebo product maltodextrin:equal amounts of a digestible carbohydrate.

Primary endpoints are faecal microbiota analysis and faecal metabolite analysis (particularly, short chain fatty acid). Secondary endpoint is serum cholesterol, glucose, HDL and bowel function, gastrointestinal tolerance, quality of life and food frequency (by the use of questionnaires).

DETAILED DESCRIPTION:
Participants will be identified and recruited at the HNU and RIHN. Participants will be informed about the study aims and procedures and will be pre-screened on the basis of inclusion/exclusion criteria. If eligible, they will sign the informed consent and enter the study with visit 0 where a clinical and biochemical evaluation of the health status will be performed. If subjects are still eligible for the study according to all the exclusion criteria, they will be included into the trial and randomised to receive the active supplementation or placebo at visit 1 (day 5). Volunteers will be invited to commence the study in batches of 5 people.

Following 5 days of maintenance diet (their usual diet), on visit 1 (day 5) volunteers would bring their fresh faecal sample to HNU, blood sample and blood pressure measurement will be taken during their visit. The placebo or fibre supplements will be given to them, enough for the next 5 days. On visit 2 (day 10), volunteers would come to HNU to deliver their faecal sample and the next 5 days' worth of placebo or fibre supplements will be provided. Volunteers will return to HNU for visit 3 (day 15) to deliver their faecal sample, blood sample and blood pressure measurement will be taken on site. There will be a wash out period of 5 days with no study product provided to the volunteers. On visit 4 (day 20), the study intervention would then cross-over and the volunteers will deliver their faecal sample to HNU. Blood sample and blood pressure measurement will be taken and the volunteers will be given the next set of products, enough for the next 5 days. On visit 5 (day 25), volunteers would come to HNU to deliver their faecal sample and the next 5 days' worth of placebo or fibre supplement will be given to them. At the end of the second intervention (day 30), volunteers will come in for visit 6 to deliver their faecal sample and have blood sample and blood pressure measurement taken.

The study will end with 5 days of wash out period, where volunteers consume their own usual diet. Volunteers would come to HNU for a final visit 7 (day 35), faecal sample will be collected at the end of the wash out period.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 60 years and above
* Body mass index 20-32 kg/m2

Exclusion Criteria:

* Fructose intolerance/ or any of the ingredients in the prebiotic mix
* On prescription antibiotics within the past 3 months
* Bowel disorder
* Vegetarian or vegan
* Eating disorders and food intolerances (restricted eating)
* Wheat and gluten allergy, coeliac disease
* Alcohol and/or other substance abuse
* Regular intake of prebiotic or probiotic supplements
* Smoking
* Psychiatric disorders resulting in perceived inability to give informed consent (including severe depression, lithium treatment, schizophrenia, severe behavioural disorders)
* Lipid/Cholesterol lowering medication (as cholesterol is one of the endpoints of the study)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Changes in the gut microbiota metabolites | Faecal samples collected on each test day (day 5, 10, 15, 20, 25, 30, 35) over an expected period of 35 days
  Samples will be used for metabolite analysis using short chain fatty acid analysis.

SECONDARY OUTCOMES:
Changes in the gut microbiota | Faecal samples collected on each test day (day 5, 10, 15, 20, 25, 30, 35) over an expected period of 35 days
  Sample will be used for microbiota analysis using molecular methods such as high-throughput sequencing and qPCR.
Changes in blood glucose | Blood samples collected on test visit 1, 3, 4, 6 (day 5, 15, 20, 30) over an expected period of 35 days
  Blood samples will be measured for glucose using the Cholestech method.
Changes in blood HDL | Blood samples collected on test visit 1, 3, 4, 6 (day 5, 15, 20, 30) over an expected period of 35 days
  Blood samples will be measured for HDL using the Cholestech method.
Changes in blood LDL | Blood samples collected on test visit 1, 3, 4, 6 (day 5, 15, 20, 30) over an expected period of 35 days
  Blood samples will be measured for LDL using the Cholestech method.
Changes in blood triglycerides | Blood samples collected on test visit 1, 3, 4, 6 (day 5, 15, 20, 30) over an expected period of 35 days
  Blood samples will be measured for triglycerides using the Cholestech method.
Changes in blood cholesterol | Blood samples collected on test visit 1, 3, 4, 6 (day 5, 15, 20, 30) over an expected period of 35 days
  Blood samples will be measured for cholesterol using the Cholestech method.
Gastrointestinal tolerance | This is assessed via a daily questionnaire throughout the whole study period of 35 days.
  A daily questionnaire will be asked on:
  * Nausea
  * Bloating
  * Flatulence
  * Cramps
  * Bowel movements
  * Stool appearance
Volunteer's habitual diet food intake | This is assessed via questionnaires given at the start and end of the study (day 0 and day 35)
  A Food Frequency Questionnaire (FFQ) will be completed at the start and the end of the study. http://www.foodfrequency.org/
General health and well-being (This is assessed via questionnaires at the end of the study) | day 35
  A health survey will be completed at the end of the study on activities, physical and emotional well-being.
Changes in faecal inflammatory markers | Faecal samples collected on each test day (day 5, 10, 15, 20, 25, 30, 35) over an expected period of 35 days
  Faecal calprotectin will be measured using ELISA method.

CONTACTS AND LOCATIONS:
Overall Officials: Harry J Flint, Professor, Principal Investigator — Rowett Institute of Nutrition and Health, University of Aberdeen
Locations (1):
- Rowett Institute of Nutrition and Health, University of Aberdeen, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Claesson MJ, Jeffery IB, Conde S, Power SE, O'Connor EM, Cusack S, Harris HM, Coakley M, Lakshminarayanan B, O'Sullivan O, Fitzgerald GF, Deane J, O'Connor M, Harnedy N, O'Connor K, O'Mahony D, van Sinderen D, Wallace M, Brennan L, Stanton C, Marchesi JR, Fitzgerald AP, Shanahan F, Hill C, Ross RP, O'Toole PW. Gut microbiota composition correlates with diet and health in the elderly. Nature. 2012 Aug 9;488(7410):178-84. doi: 10.1038/nature11319. PMID 22797518
- [Background] Cloetens L, Broekaert WF, Delaedt Y, Ollevier F, Courtin CM, Delcour JA, Rutgeerts P, Verbeke K. Tolerance of arabinoxylan-oligosaccharides and their prebiotic activity in healthy subjects: a randomised, placebo-controlled cross-over study. Br J Nutr. 2010 Mar;103(5):703-13. doi: 10.1017/S0007114509992248. Epub 2009 Dec 10. PMID 20003568
- [Background] Duncan SH, Hold GL, Harmsen HJM, Stewart CS, Flint HJ. Growth requirements and fermentation products of Fusobacterium prausnitzii, and a proposal to reclassify it as Faecalibacterium prausnitzii gen. nov., comb. nov. Int J Syst Evol Microbiol. 2002 Nov;52(Pt 6):2141-2146. doi: 10.1099/00207713-52-6-2141. PMID 12508881
- [Background] Duncan SH, Flint HJ. Probiotics and prebiotics and health in ageing populations. Maturitas. 2013 May;75(1):44-50. doi: 10.1016/j.maturitas.2013.02.004. Epub 2013 Mar 11. PMID 23489554
- [Background] Flint HJ, Scott KP, Louis P, Duncan SH. The role of the gut microbiota in nutrition and health. Nat Rev Gastroenterol Hepatol. 2012 Sep 4;9(10):577-89. doi: 10.1038/nrgastro.2012.156. eCollection 2012 Oct. PMID 22945443
- [Background] Francois IE, Lescroart O, Veraverbeke WS, Marzorati M, Possemiers S, Evenepoel P, Hamer H, Houben E, Windey K, Welling GW, Delcour JA, Courtin CM, Verbeke K, Broekaert WF. Effects of a wheat bran extract containing arabinoxylan oligosaccharides on gastrointestinal health parameters in healthy adult human volunteers: a double-blind, randomised, placebo-controlled, cross-over trial. Br J Nutr. 2012 Dec 28;108(12):2229-42. doi: 10.1017/S0007114512000372. Epub 2012 Feb 28. PMID 22370444
- [Background] Francois IE, Lescroart O, Veraverbeke WS, Marzorati M, Possemiers S, Hamer H, Windey K, Welling GW, Delcour JA, Courtin CM, Verbeke K, Broekaert WF. Effects of wheat bran extract containing arabinoxylan oligosaccharides on gastrointestinal parameters in healthy preadolescent children. J Pediatr Gastroenterol Nutr. 2014 May;58(5):647-53. doi: 10.1097/MPG.0000000000000285. PMID 24368315
- [Background] Hopkins MJ, Sharp R, Macfarlane GT. Age and disease related changes in intestinal bacterial populations assessed by cell culture, 16S rRNA abundance, and community cellular fatty acid profiles. Gut. 2001 Feb;48(2):198-205. doi: 10.1136/gut.48.2.198. PMID 11156640
- [Background] Lewis SJ, Heaton KW. Increasing butyrate concentration in the distal colon by accelerating intestinal transit. Gut. 1997 Aug;41(2):245-51. doi: 10.1136/gut.41.2.245. PMID 9301506
- [Background] Maki KC, Gibson GR, Dickmann RS, Kendall CW, Chen CY, Costabile A, Comelli EM, McKay DL, Almeida NG, Jenkins D, Zello GA, Blumberg JB. Digestive and physiologic effects of a wheat bran extract, arabino-xylan-oligosaccharide, in breakfast cereal. Nutrition. 2012 Nov-Dec;28(11-12):1115-21. doi: 10.1016/j.nut.2012.02.010. Epub 2012 Jul 6. PMID 22771050
- [Background] Maloy KJ, Powrie F. Intestinal homeostasis and its breakdown in inflammatory bowel disease. Nature. 2011 Jun 15;474(7351):298-306. doi: 10.1038/nature10208. PMID 21677746
- [Background] Parracho H, McCartney AL, Gibson GR. Probiotics and prebiotics in infant nutrition. Proc Nutr Soc. 2007 Aug;66(3):405-11. doi: 10.1017/S0029665107005678. PMID 17637093
- [Background] Pryde SE, Duncan SH, Hold GL, Stewart CS, Flint HJ. The microbiology of butyrate formation in the human colon. FEMS Microbiol Lett. 2002 Dec 17;217(2):133-9. doi: 10.1111/j.1574-6968.2002.tb11467.x. PMID 12480096
- [Background] Rastall RA, Maitin V. Prebiotics and synbiotics: towards the next generation. Curr Opin Biotechnol. 2002 Oct;13(5):490-6. doi: 10.1016/s0958-1669(02)00365-8. PMID 12459343
- [Background] Scott KP, Gratz SW, Sheridan PO, Flint HJ, Duncan SH. The influence of diet on the gut microbiota. Pharmacol Res. 2013 Mar;69(1):52-60. doi: 10.1016/j.phrs.2012.10.020. Epub 2012 Nov 9. PMID 23147033
- [Background] Sokol H, Pigneur B, Watterlot L, Lakhdari O, Bermudez-Humaran LG, Gratadoux JJ, Blugeon S, Bridonneau C, Furet JP, Corthier G, Grangette C, Vasquez N, Pochart P, Trugnan G, Thomas G, Blottiere HM, Dore J, Marteau P, Seksik P, Langella P. Faecalibacterium prausnitzii is an anti-inflammatory commensal bacterium identified by gut microbiota analysis of Crohn disease patients. Proc Natl Acad Sci U S A. 2008 Oct 28;105(43):16731-6. doi: 10.1073/pnas.0804812105. Epub 2008 Oct 20. PMID 18936492
- [Background] Suau A, Bonnet R, Sutren M, Godon JJ, Gibson GR, Collins MD, Dore J. Direct analysis of genes encoding 16S rRNA from complex communities reveals many novel molecular species within the human gut. Appl Environ Microbiol. 1999 Nov;65(11):4799-807. doi: 10.1128/AEM.65.11.4799-4807.1999. PMID 10543789
- [Background] Walker AW, Ince J, Duncan SH, Webster LM, Holtrop G, Ze X, Brown D, Stares MD, Scott P, Bergerat A, Louis P, McIntosh F, Johnstone AM, Lobley GE, Parkhill J, Flint HJ. Dominant and diet-responsive groups of bacteria within the human colonic microbiota. ISME J. 2011 Feb;5(2):220-30. doi: 10.1038/ismej.2010.118. Epub 2010 Aug 5. PMID 20686513
- [Background] Zheng G, Yampara-Iquise H, Jones JE, Andrew Carson C. Development of Faecalibacterium 16S rRNA gene marker for identification of human faeces. J Appl Microbiol. 2009 Feb;106(2):634-41. doi: 10.1111/j.1365-2672.2008.04037.x. PMID 19200327
- [Derived] Chung WSF, Walker AW, Bosscher D, Garcia-Campayo V, Wagner J, Parkhill J, Duncan SH, Flint HJ. Relative abundance of the Prevotella genus within the human gut microbiota of elderly volunteers determines the inter-individual responses to dietary supplementation with wheat bran arabinoxylan-oligosaccharides. BMC Microbiol. 2020 Sep 14;20(1):283. doi: 10.1186/s12866-020-01968-4. PMID 32928123